CLINICAL TRIAL: NCT02892292
Title: Next Generation Sequencing (NGS) Application for HLA Typing of Donors and Recipients of Hematopoietic Stem Cells
Brief Title: NGS for HLA Typing of Donors and récipients oh Hematopoietic Stem Cells
Acronym: NGS HLA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: NGS-HLA
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Next Generation Sequencing for HLA Typing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to realize the typing of all HLA loci and validate this technique with continued optimization of next-generation sequencing technology (NGS).

DETAILED DESCRIPTION:
The number of patients waiting allograft of hematopoietic stem cells is constantly evolving. Similarly, the number of voluntary donors of hematopoietic stem cells on all global file has exceeded the threshold of 22 million donors since the end of 2013. Despite this, the search for a matched unrelated donor HLA for a patient remains sometimes a long and difficult, especially for patients with rare HLA alleles. It is important to increase the number of donors in the global file, increase HLA diversity of registrants and resolution HLA typing. More HLA typing of a donor registered on the file will be accurate, more research and the recruitment of a donor in order to achieve an allograft in a patient waiting will be fast.

The constant evolution of the number of HLA alleles and the number of ambiguities quickly demonstrates the limits of current typing techniques. The study of exons and introns that would significantly refine the level of resolution HLA typing, reaching a level of allelic resolution. That level of resolution would also identify all null alleles (alleles from which the protein is not expressed). The search for an HLA with a patient will be made easier by reducing the financial impact and time of the search. In addition, numerous studies have shown that tissue compatibility narrowest possible between the donor and recipient of an allogeneic haematopoietic stem cells can improve patient survival by reducing the incidence and severity of disease graft against the host and to improve engraftment.

In addition, analysis capability of the many sample using this technique should induce the decrease in HLA typing costs and thus facilitate the registration of anonymous bone marrow donors on the national register of the Biomedicine Agency .

ELIGIBILITY:
Inclusion Criteria:

* Bone marrow donors from Brest University Hospital
* Bone marrow recipients of Brest University Hospital

Exclusion Criteria:

* No bone marrow donors from Brest University Hospital
* No bone marrow recipients of Brest University Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bone marrow donors-recipients of Brest University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
HLA high resolution sequencing for loci HLA-A, HLA-B, HLA-C, HLA-DRB1, HLA-DQB1 and HLA-DPB1. | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Moalic-Allain, Doctor, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France